CLINICAL TRIAL: NCT00917306
Title: A Multi-center, Open-label Study to Evaluate the Safety and Efficacy of PEP005 (Ingenol Mebutate) Gel, 0.05% in Patients With Actinic Keratoses on Non-head Locations (Trunk and Extremities)
Brief Title: A Multi-center Study to Evaluate the Safety and Efficacy of PEP005 (Ingenol Mebutate) Gel, When Used to Treat Actinic Keratoses on Non-head Locations (Trunk and Extremities)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peplin (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-020
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEP005 gel (Experimental): PEP005 gel, 0.05% administered once daily for 2 consecutive days
  Interventions: Drug: PEP005 Gel

INTERVENTIONS:
Drug: PEP005 Gel — 0.05% two day treatment
  Other Names: PEP005

SUMMARY:
The open label study is designed to assess the safety and efficacy of 0.05% PEP005 Gel when applied to an area of skin containing 4-8 AK lesions on non-head locations.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and at least 18 years of age.
* Female patient must be of either:

  * Non-childbearing potential, post-menopausal, or there is a confirmed clinical history of sterility (e.g., the patient is without a uterus)
  * Childbearing potential, provided there are negative urine pregnancy test results prior to study treatment, to rule out pregnancy

Exclusion Criteria

* Cosmetic or therapeutic procedures within two weeks and within 2 cm of the selected treatment area.
* Treatment with immunomodulators, interferon/ interferon inducers or systemic medications that suppress the immune system within 4 weeks.
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 8 weeks and 2 cm of the selected treatment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety (Incidence of treatment related AEs, local skin reactions and pigmentation and scarring) | 57 days

SECONDARY OUTCOMES:
Efficacy (complete and partial clearance of AK lesions) | 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Bauer, MD, Study Director — Chief Medical Officer
Locations (11):
- United States (8):
  - Park Avenue Dermatology, Orange Park, Florida
  - Medaphase Inc, Newnan, Georgia
  - Gwinnett Clinical Research Centre, Snellville, Georgia
  - Michigan Center for Research Corp, Clinton Twp, Michigan
  - Henry Ford Health Systems, Detroit, Michigan
  - Dermatology Associates of Rochester, Rochester, New York
  - Oregon Health and Science University, Portland, Oregon
  - Dermatology Research Associates, Nashville, Tennessee
- Australia (3):
  - Dematology on Ward, Adelaide, South Australia
  - Dermatology Institute of Victoria, Melbourne, Victoria
  - St John of God Dermatology, Subiaco, Western Australia

REFERENCES:
- See also: Food and Drug Authority — http://www.fda.gov
- See also: Therapeutic Goods Administration — http://tga.gov.au